CLINICAL TRIAL: NCT02850666
Title: Building Social Skills in Children With ASD Characteristics Through Process Drama
Brief Title: Social Skills in Children With ASD and Process Drama
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Lorie Richards, Chair and Associate Professor, University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB_00091961
Record Dates: First submitted 2016-07-26; First posted 2016-08-01 (Estimated); Last update posted 2018-05-15 (Actual); Status verified 2018-05

CONDITIONS: Autistic Disorder
Keywords: social skills; child; theory of mind; drama; occupational therapy; Speech-language pathology
MeSH Terms: conditions — Autistic Disorder; Social Skills

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Interdisciplinary Process drama (Experimental): Process drama program (5 days/week, 1 week, 25-3 hour sessions) of movement-based activities combining music, art, and drama. Activities have been planned by a collaborative team of drama teachers, occupational therapists, and speech language pathologists.
  Interventions: Behavioral: Interdisciplinary process drama

INTERVENTIONS:
Behavioral: Interdisciplinary process drama — Process drama program (5 days/week, 1 week, 25-3 hour sessions) of movement-based activities combining music, art, and drama. Activities have been planned by a collaborative team of drama teachers, occupational therapists, and speech language pathologists.

SUMMARY:
This is a one-group, pre-post feasibility study of an intensive, interdisciplinary (theatre, Occupational Therapy (OT), and Speech Language Pathology (SLP)) intervention targeted at social skill development in children, aged 3-4. The intervention uses process drama modified with OT and SLP techniques and using typically developing peer models. Feasibility outcomes are recruitment rates, retention rates, daily program records of ease of implementing program, and record of modifications needed. Child primary outcomes are Social Skills Improvement Scale (SSIS), Theory of Mind (T0M) Battery and Inventory, Structured Play Assessment (SPA), and Communication and Symbolic Behavior Scales (CSBS) scores within 4 weeks of program end. Secondary outcomes are brain activity in frontal lobe and temporal/parietal areas measured by high density EEG within 4 weeks of program end, parental interview at 3 months related to child's social skills, and observational data on social skills during the program.

DETAILED DESCRIPTION:
Six children with Autism Spectrum Disorder (ASD) and 6 typically developing (TD) preschool children participate will complete baseline testing. The TD children will only complete the EEG testing, while the ASD children and their parents will complete all outcome assessments. In addition to the outcome measures listed in the Brief Summary, the children we will administer the the Vineland Adaptive Behavioral Scales (Vineland - II), the Mullen Scales of Early Learning, and the Autism Diagnostic Observation Scale - II (if they have not had one administered within the past 12 months) for sample description.

During the EEG session, brain activity during theory of mind and other social stimuli will be used to measure brain behavior relationships. The recordings will adhere to standard clinical EEG procedures, using high density EEG providing a high spatial resolution for electrical source imaging in brain space. They will be conducted by a Registered EEG Technologist (R. EEG T) with a specially trained student assistant. The procedure will involve first explaining to the parent and child what will be done. The participants will sit within a chair or a parent's lap while the EEG is recorded. The EEG tasks will consist of the following: First the child will be asked to open and close their eyes for a few minutes to record a baseline resting EEG. Then there will be both auditory sounds (intonations and word components) and images of social stimuli embedded between fun cartoon stimuli to maintain the child's attention displayed on a screen. The pictures will consist of eye movements, facial gestures, and point light diagrams of body movements.

The process drama program will be conducted with 6 children with ASD and 6 TD peer models 5 days per week for 1 week for 2.5-3 hours each day. The program will consist of several sections. Each day will open with an opening ritual that is movement based involving mirroring activity. This is followed by a welcome/greeting activity, involving things like a song and Name activity. The remainder of the activities build around a story for the day. The story will be one that holds interest for young children, such as a day in the life of a tree who gets visited by animals and people. The story unfolds with problems to solve and social interactions to do. Participants and the drama teachers take on different roles to bring out the story. Engagement starts out with drama pieces that the children can do individually and progress to those requiring a partner and then small groups. Other artistic experiences related to the story are included in the session, such as music and movement related to the story and an art activity related to the story. The sessions close with a closing ritual, reminding the participants of what was done during the session and a song. All the activities focus on building understanding the emotions and intentions of others and appropriate social interactions. The setting of the program and the specific activities have been planned with a collaborative team of drama teachers, an occupational therapists, and a speech language pathologists.

The process drama sessions will be videotaped and later scored for social interactions and social verbal and non-verbal communication. We will also examine the engagement of the participants with ASD to determine if we need to change/alter any procedures/techniques that we are using during the process drama sessions in subsequent versions of this research. We will also examine the behavior of the peer models to identify areas in which the research team may need to change to better engage the peer models in subsequent sessions.

After the end of the process drama intervention, the participants with ASD will repeat the baseline assessments within 4 weeks of intervention end. The assessments that will be repeated are the ToMT, CSBS, SPA and SSiS. The children with ASD will also complete another EEG session as they did at baseline.

Three months after the last testing session, the parents will be contacted to complete an interview to ask how their children are functioning related to play and other interactions with other children and with adults. These interviews may occur face-to-face at a mutually agreed upon location, could be over the phone, or could be via a video conferencing system, such as Business Skype. The interviews will be audio-recorded for later thematic analysis. After these themes are identified, the parents will be re-contacted and shown the identified themes to make sure that we have accurately represented what they intended to convey (member checking).

ELIGIBILITY:
Inclusion Criteria: Participants with ASD:

* aged 3-4 years old
* documented diagnosis of ASD from a licensed professional using DSM 5 criteria12; If no documentation available, meets cut off on Autism Diagnostic Observation Scale (ADOS -2)13 that will be administered by trained study staff.
* passes language and cognitive screen (see attached screening document with decision rules) and a receptive language age equivalence of ≥18 months and a non-verbal age equivalent score of ≥24 months on the Mullen Scale of Early Learning14
* have a caregiver willing/able to bring them to the University for the study sessions and to schedule up to 3 assessment visits prior to intervention start and 3 assessment sessions after intervention end
* family's primary language is English

Typically developing children

* aged 3-4
* normal or corrected to normal vision and hearing
* English speaking

Exclusion Criteria: Participants with ASD

* have no other major medical conditions (i.e., no genetic disorders such as Fragile X, Down syndrome)
* seizure disorder
* uncorrected hearing or visual impairment
* other condition causing motor impairment, such as Cerebal Palsy

Typically developing children

-no history of developmental delay or neurological disorder

Ages: 3 Years to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 11 (Actual)
Dates: Start 2016-07; Primary Completion 2017-09-12 (Actual); Study Completion 2017-10-01 (Actual)

PRIMARY OUTCOMES:
Social Skills Improvement Scale | 4 weeks post intervention
  Child primary outcome: Parent rating of statements about child's social interactions
Theory of Mind Battery and Inventory | 4 weeks post intervention
  Child primary outcome: performance test of theory of mind activities and parent ratings of statements of child behavior in theory of mind situations
Structured Play Assessment | 4 weeks after intervention
  Performance test of how child plays with toys
Retention Rate | 3 months after intervenrtion
  Feasibility outcome: number of participants who completed 4 week assessments and 3 month parent interview
Recruitment | at baseline
  ability to recruit needed number of participants in time frame availability

SECONDARY OUTCOMES:
Brain activity during Theory of Mind tasks | 4 weeks after intervention
  Dense EEG recordings of brain activity in frontal/temporal/and parietal lobes during TOM tasks
Parental perceptions of social skills | 3 months
  Interview with parent regarding changes seen in social skills
Changes in social skills during program | 1 week
  observations (via video recording) of social skills during intervention program
Modifications needed to program | at 1 week
  record of modifications made during the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Lorie G Richards, PhD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pelphrey KA, Morris JP, McCarthy G. Grasping the intentions of others: the perceived intentionality of an action influences activity in the superior temporal sulcus during social perception. J Cogn Neurosci. 2004 Dec;16(10):1706-16. doi: 10.1162/0898929042947900. PMID 15701223
- [Background] Thomas MS, Davis R, Karmiloff-Smith A, Knowland VC, Charman T. The over-pruning hypothesis of autism. Dev Sci. 2016 Mar;19(2):284-305. doi: 10.1111/desc.12303. Epub 2015 Apr 6. PMID 25845529
- [Result] Corbett BA, Key AP, Qualls L, Fecteau S, Newsom C, Coke C, Yoder P. Improvement in Social Competence Using a Randomized Trial of a Theatre Intervention for Children with Autism Spectrum Disorder. J Autism Dev Disord. 2016 Feb;46(2):658-72. doi: 10.1007/s10803-015-2600-9. PMID 26419766